CLINICAL TRIAL: NCT03921671
Title: Improving Treatment Strategies in Thymic Epithelial Tumors: a TYME Collaborative Effort
Brief Title: Ramucirumab and Carbo-Paclitaxel for Untreated Thymic Carcinoma / B3 Thymoma With Carcinoma (RELEVENT)
Acronym: RELEVENT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Claudia Proto (Other)
Responsible Party: Sponsor-Investigator, Claudia Proto, Principal Investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Organization: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-TET1-7371; 2017-004494-13 (EudraCT Number)
Record Dates: First submitted 2018-06-22; First posted 2019-04-19 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-02

CONDITIONS: Thymic Carcinoma; Thymoma
Keywords: metastatic or relapsed non-pre-treated disease
MeSH Terms: conditions — Thymoma; Neoplasm Metastasis | interventions — Ramucirumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Green-Dahlberg 2-stage design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ramucirumab +carboplatin+ paclitaxel (Experimental): All patient will receive the combination of ramucirumab (10 mg / kg) + carboplatin (AUC 5) and paclitaxel (200 mg / m2) in patients with recurrent and / or metastatic thymic carcinoma or thymoma B3 with area of carcinoma, in the first line.
  Interventions: Combination Product: Ramucirumab

INTERVENTIONS:
Combination Product: Ramucirumab — Combination of ramucirumab (10 mg / kg) + carboplatin (AUC 5) and paclitaxel (200 mg / m2) in patients with carcinoma thymic (or thymoma B3 with areas of carcinoma), relapsed and / or metastatic, in the first line.
  Other Names: CARBOPLATIN (AUC 5) + PACLITAXEL(200 mg / m2)

SUMMARY:
This is a multicentric study. All patients with TET (thymic epithelial tumors) of any histological type will participate in the study. This is an open-label phase 2 study that will follow a Green-Dahlberg 2-stage design whose objective is to evaluate the activity and safety of the combination of ramucirumab (10 mg / kg) + carboplatin (AUC 5) and paclitaxel (200 mg / m2) in patients with relapsed and / or metastatic thymic carcinoma/ thymoma B3, in the first line (RELEVENT trial).

DETAILED DESCRIPTION:
Clinical and quality of life data will be collected for all treated patient. Based on the histological evaluation performed by each participating center, patients will be screened for inclusion in one of the four studies, based on the following criteria:

* TOPS study only: all patients with A, AB, B1, B2, B3 without areas of carcinoma histology, diagnosed during or after 2018, that do not have a fresh tissue sample and screen failures of the RELEVENT and BIOTET study;
* TRY registry: all patients with TETs diagnosed, treated or followed from 2010 to 2017 included (retrospective data collection);
* BIOTET only: all patients with A, AB, B1, B2, B3 without areas of histology of the carcinoma that have a fresh tissue sample;
* RELEVENT only: all patients with thymoma B3 and areas of carcinoma and pa-tients with thymic carcinoma who do not have a fresh tissue sample.

Patients with thymic carcinoma or thymoma B3 with areas of carcinoma will receive a centralized pathological review of the tumour block or slides and will be screened to participate in the Phase II RELEVENT pharmacological study.Histological diagnosis will be confirmed before screening.

ELIGIBILITY:
Inclusion Criteria:

1. provision of written informed consent before treatment initiation
2. pathologically confirmed thymic carcinoma and B3 thymomas, with areas of carcinoma locally advanced as per central histological revision, recurrent and/or metastatic, not amenable to potentially curative treatments.
3. age>= 18 years old
4. provision of archival or fresh tissue (block or at least 15 charged slides 4μM of thickness).
5. Blood and plasma sampling at baseline and at first clinical revaluation
6. measurable disease (defined according to Response Evaluation Criteria in Solid Tumours [RECIST] version 1.1);7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;

8. adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥1500/μL, haemoglobin

≥9 g/dL (5.58 mmol/L), and platelets ≥100,000/μL; 9. adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Patients receiving warfarin must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to first dose of protocol therapy 10. adequate hepatic function as defined by a total bilirubin ≤1.5times the upper limit of normal (ULN), (Except for patients with Gilbert's syndrome who may only be included in the total bilirubin is < 3.0 x ULN or direct bilirubin < 1.5 x ULN) and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 times the upper limit of normal (or 5.0 times the ULN in the setting of liver metastases) 11. adequate renal function as defined by a serum creatinine ≤1.5 times the ULN, or creatinine clearance (measured via 24-hour urine collection) ≥40 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed). The patient's urinary protein is

≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol).

12. sexually active patients, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods). Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to first dose of protocol therapy. 13. Prior radiation therapy is allowed.

* In case of chest radiotherapy a 28 days interval is needed between the end of the radiation treatment and the start of treatment .
* In the case of focal or palliative radiation treatment a 7 days interval is needed from last radiation treatment to start of treatment (and provided that 25% or less of total bone marrow had been irradiated).
* In the case of CNS radiation a minimum of 14 days interval is needed from the end of radiation treatment to start of treatment.

Exclusion Criteria:

1. previous systemic treatment for locally advanced/metastatic thymic carcinoma/B3 thymomas; patients treated in the neoadjuvant or adjuvant setting can be enrolled after discussion with PI
2. untreated CNS metastases. Patients with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, and stereotactic radiosurgery) ending at least 2 weeks prior to start of treatment, or after surgical resection performed at least 28 days prior to start of treatment. The patient may have no evidence of Grade ≥1 CNS haemorrhage based on pre-treatment Magnetic Resonance Imaging (MRI) or IV contrast CT scan (performed within 28 days before start of treatment)
3. any Grade 3-4 GI bleeding within 3 months prior to first dose of protocol therapy
4. peripheral neuropathy ≥ G2History of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy.
5. patient has experienced hemoptysis (defined as bright red blood or ≥ 1/2 teaspoon) within 2 months prior to first dose of protocol therapy
6. radiographic evidence of intra-tumour cavitation, radiologically documented evidence of major blood vessel invasion or encasement by cancer
7. history of uncontrolled hereditary or acquired thrombotic disorder
8. The patient has:

   * cirrhosis at a level of Child-Pugh B (or worse) or
   * cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis.
9. clinically relevant congestive heart failure (NYHA II-IV) or symptomatic or poorly controlled cardiac arrhythmia
10. The patient has experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to first dose of protocol therapy.uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management.
11. serious or no healing wound, ulcer, or bone fracture within 28 days prior to start of treatment
12. significant bleeding disorders, vasculitis, or experienced grade 3/4 gastrointestinal (GI) bleeding within 3 months prior to start of treatment
13. history of GI perforation and / or fistulae within 6 months prior to start of treatment
14. bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection, Crohn's disease, ulcerative colitis, or chronic diarrhoea
15. peripheral neuropathy ≥grade 2 (NCI-CTCAE v 4.0)
16. serious illness or medical condition(s) including, but not limited to, the following: -Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)- related illness.

    * Active or uncontrolled clinically serious infection.
    * Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumours treated curatively and without evidence of recurrence for at least 3 years prior to start of treatment.
    * Uncontrolled metabolic disorders or other non-malignant organ or systemic diseases or secondary effects of cancer that induce a high medical risk and/or make assessment of survival uncertain.
    * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient ineligible for entry into this study.
    * significant third-space fluid retention (for example, ascites or pleural effusion), and is not amenable for required repeated drainage
17. known allergy or hypersensitivity reaction to any of the treatment components
18. known history of active drug abuse
19. patient is pregnant or breastfeeding
20. major surgery within 28 days prior to first dose of protocol therapy, or minor surgery/subcutaneous venous access device placement within 7 days prior to first dose of protocol therapy
21. elective or planned major surgery to be performed during the course of the clinical trial
22. patient is receiving concurrent treatment with other anticancer therapy
23. patient is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents.

Once-daily aspirin use (maximum dose 325 mg/day) is permitted.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2024-07-16 (Estimated)

PRIMARY OUTCOMES:
Best tumour response (CR+PR) | 6 months
  Objective tumor response will be assessed according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 4 years
  Disease progression will be established as the radiological progression according to RECIST 1.1 or through clinical assessment in case radiological evaluation is not feasible or as death from any cause due to clinical condition. PFS will be estimated through Kaplan-Meier method
Overall Survival (OS) | 4 years
  OS will be estimated through Kaplan-Meier method
Safety | 4 years
  AE/SAE will be reported and graded. Evaluaton of relationship with experimental drug will be done

OTHER OUTCOMES:
Comprehensive analysis of tumor mutational status on paraffin-embedded tissue | 4 years
  Targeted re-sequencing of genes mutated in TETs in order to define the prognostic role of somatic mutations and their potential association to prognosis or response to therapy
Comprehensive analysis of single nucleotide polymorphism in blood | 4 years
  Genome-wide approach using a platform able to investigate more than 4 million SNP in order to find potential association with prognosis or response to therapy
Analysis of circulating micro-RNA | 4 years
  Analysis of micro-RNA in plasma and their evaluation as possible biomarker associated with prognosis or response to therapy
Quality of life analysis through collection of Patients Reported Outcome (PROs) | 4 years
  Web based PROs will be administered at each visit and data about compliance will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Marina Garassino, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
hospital records; clinical and office charts, laboratory and pharmacy records, diaries, microfiches, radiographs, and correspondence. Data collection will be performed using electronic CRFs exclusively. No paper CRFs are provided to study investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the first patient enrolled, to the end of the study
Access Criteria: Direct access to source data will be granted to authorised representatives from the Sponsor, host institution and the regulatory authorities to permit trial-related monitoring, audits and inspections.
  Access to the study clinical data entry platform will be granted to trial staff through a computer-based credential generation system in the following manner:

REFERENCES:
- [Result] Benveniste MF, Korst RJ, Rajan A, Detterbeck FC, Marom EM; International Thymic Malignancy Interest Group. A practical guide from the International Thymic Malignancy Interest Group (ITMIG) regarding the radiographic assessment of treatment response of thymic epithelial tumors using modified RECIST criteria. J Thorac Oncol. 2014 Sep;9(9 Suppl 2):S119-24. doi: 10.1097/JTO.0000000000000296. PMID 25396308
- [Result] Berruti A, Borasio P, Gerbino A, Gorzegno G, Moschini T, Tampellini M, Ardissone F, Brizzi MP, Dolcetti A, Dogliotti L. Primary chemotherapy with adriamycin, cisplatin, vincristine and cyclophosphamide in locally advanced thymomas: a single institution experience. Br J Cancer. 1999 Nov;81(5):841-5. doi: 10.1038/sj.bjc.6690773. PMID 10555755
- [Result] Enkner F, Pichlhofer B, Zaharie AT, Krunic M, Holper TM, Janik S, Moser B, Schlangen K, Neudert B, Walter K, Migschitz B, Mullauer L. Molecular Profiling of Thymoma and Thymic Carcinoma: Genetic Differences and Potential Novel Therapeutic Targets. Pathol Oncol Res. 2017 Jul;23(3):551-564. doi: 10.1007/s12253-016-0144-8. Epub 2016 Nov 14. PMID 27844328
- [Result] Garg RK. Posterior leukoencephalopathy syndrome. Postgrad Med J. 2001 Jan;77(903):24-8. doi: 10.1136/pmj.77.903.24. PMID 11123390
- [Result] Lopez-Garcia F, Amoros-Martinez F, Sempere AP. [A reversible posterior leukoencephalopathy syndrome]. Rev Neurol. 2004 Feb 1-15;38(3):261-6. Spanish. PMID 14963856
- [Result] Hirai F, Yamanaka T, Taguchi K, Daga H, Ono A, Tanaka K, Kogure Y, Shimizu J, Kimura T, Fukuoka J, Iwamoto Y, Sasaki H, Takeda K, Seto T, Ichinose Y, Nakagawa K, Nakanishi Y; West Japan Oncology Group. A multicenter phase II study of carboplatin and paclitaxel for advanced thymic carcinoma: WJOG4207L. Ann Oncol. 2015 Feb;26(2):363-8. doi: 10.1093/annonc/mdu541. Epub 2014 Nov 17. PMID 25403584
- [Result] Hesketh PJ, Kris MG, Basch E, Bohlke K, Barbour SY, Clark-Snow RA, Danso MA, Dennis K, Dupuis LL, Dusetzina SB, Eng C, Feyer PC, Jordan K, Noonan K, Sparacio D, Somerfield MR, Lyman GH. Antiemetics: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2017 Oct 1;35(28):3240-3261. doi: 10.1200/JCO.2017.74.4789. Epub 2017 Jul 31. PMID 28759346
- [Result] Lee VH, Wijdicks EF, Manno EM, Rabinstein AA. Clinical spectrum of reversible posterior leukoencephalopathy syndrome. Arch Neurol. 2008 Feb;65(2):205-10. doi: 10.1001/archneurol.2007.46. PMID 18268188
- [Result] Lemma GL, Lee JW, Aisner SC, Langer CJ, Tester WJ, Johnson DH, Loehrer PJ Sr. Phase II study of carboplatin and paclitaxel in advanced thymoma and thymic carcinoma. J Clin Oncol. 2011 May 20;29(15):2060-5. doi: 10.1200/JCO.2010.32.9607. Epub 2011 Apr 18. PMID 21502559
- [Result] Marinella MA, Markert RJ. Reversible posterior leucoencephalopathy syndrome associated with anticancer drugs. Intern Med J. 2009 Dec;39(12):826-34. doi: 10.1111/j.1445-5994.2008.01829.x. Epub 2008 Nov 3. PMID 19220526
- [Result] Okuma Y, Saito M, Hosomi Y, Sakuyama T, Okamura T. Key components of chemotherapy for thymic malignancies: a systematic review and pooled analysis for anthracycline-, carboplatin- or cisplatin-based chemotherapy. J Cancer Res Clin Oncol. 2015 Feb;141(2):323-31. doi: 10.1007/s00432-014-1800-6. Epub 2014 Aug 22. PMID 25146529
- [Result] Pagano M, Sierra NM, Panebianco M, Rossi G, Gnoni R, Bisagni G, Boni C. Sorafenib efficacy in thymic carcinomas seems not to require c-KIT or PDGFR-alpha mutations. Anticancer Res. 2014 Sep;34(9):5105-10. PMID 25202099
- [Result] Schwartz RB. A reversible posterior leukoencephalopathy syndrome. N Engl J Med. 1996 Jun 27;334(26):1743; author reply 1746. doi: 10.1056/NEJM199606273342613. No abstract available. PMID 8637524